CLINICAL TRIAL: NCT04761939
Title: BIONICS Small Vessels Trial EluNIR Ridaforolimus Eluting Coronary Stent System (EluNIR) in Coronary Stenosis Trial
Status: Completed | Type: Observational
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EluNIR-005
Record Dates: First submitted 2020-10-11; First posted 2021-02-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Coronary Stenosis; Coronary Disease; Myocardial Ischemia; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Stenosis; Coronary Disease; Myocardial Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Combination Product: EluNIR Ridaforolimus Eluting Coronary Stent System — The EluNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising of:
  * Stent - a pre-mounted Cobalt Chromium (CoCr) alloy based stent - 2.25 mm Diameter and 8mm, 12mm, 15mm, 17mm, 20mm, 24mm, 28mm and 33mm length
  * Delivery System - Rapid Exchange (RX) Coronary System
  * Polymer matrix coating - Poly n-butyl methacrylate (PBMA) and CarboSil®
  * Ridaforolimus drug - CAS Registry Number: 572924-54-0

SUMMARY:
Device:

EluNIR Ridaforolimus Eluting Coronary Stent System - (hereafter referred to as EluNIR) 2.25 mm diameter (8 mm, 12 mm, 15 mm, 17 mm, 20 mm, 24 mm, 28 mm and 33 mm length)

Objectives:

To further assess the safety and efficacy of the small diameter (2.25 mm) Ridaforolimus Eluting Stent - EluNIR.

Subject Population:

Subjects who underwent PCI for angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present), NSTEMI, and recent STEMI (>24 hours from initial presentation and stable) with attempted implantation of a 2.25 mm diameter EluNIR stent.

Trial Design and Methods:

This is a prospective, multi-center, single-arm, open-label clinical trial. Clinical follow-up for all patients will be performed at 30 days 6 months, and 1 year after the procedure.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years. 2. Patient with an indication for PCI including angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present), NSTEMI, or recent STEMI. For STEMI the time of presentation to the first treating hospital, whether a transfer facility or the study hospital, must be >24 hours prior to enrollment and enzyme levels (CK-MB or Troponin) demonstrating that either or both enzyme levels have peaked.

3. An attempt (whether successful or not) was made to implant a 2.25 mm EluNIR stent (Stent was advanced beyond the guiding catheter).

4. Non-target lesion PCIs are allowed depending on the time interval and conditions as follows:

1. During Index Procedure:

   if successful and uncomplicated defined as: <50% visually estimated residual diameter stenosis, TIMI Grade 3 flow, no dissection ≥ NHLBI type C, no perforation, no persistent ST segment changes, no prolonged chest pain, no TIMI major or BARC type 3 bleeding.
2. Less than 24 hours prior to Index Procedure:

Not allowed (see exclusion criteria #2). c. 24 hours-30 days prior to Index Procedure: i. PCI of non-target vessels 24 hours to 30 days prior to the index procedure if successful and uncomplicated as defined above.

ii. In addition, in cases where non-target vessel PCI has occurred 24-72 hours prior to the index procedure, at least 2 sets of cardiac biomarkers must have been drawn at least 6 and 12 hours after the non-target vessel PCI.

iii. If cardiac biomarkers are initially elevated above the local laboratory upper limit of normal, serial measurements must demonstrate that the biomarkers are falling.

d. Over 30 days prior to Index Procedure: PCI of non-target lesions performed greater than 30 days prior to index procedure whether or not successful and uncomplicated.

5. Patient or legal guardian is willing and able to provide informed written consent and comply with follow-up visits and testing schedule.

Angiographic inclusion criteria (visual estimate):

6. Target lesion(s) must be located in a native coronary artery or bypass graft conduit with visually estimated diameter of ≥2.25 mm to ≤2.5 mm.

7. Complex lesions are allowed including calcified lesions (lesion preparation with scoring/cutting and rotational atherectomy are allowed), presence of thrombus, CTO, bifurcation lesions, ostial RCA lesions, tortuous lesions, bare metal stent restenotic lesions, protected left main lesions, and saphenous vein graft lesions.

8. Overlapping stents are allowed as long as at least one of the stents implanted is the EluNIR 2.25 mm diameter stent

Exclusion Criteria:

1. STEMI within 24 hours of initial time of presentation to the first treating hospital, whether at a transfer facility or the study hospital or in whom enzyme levels (either CK-MB or Troponin) have not peaked.
2. PCI within the 24 hours preceding the index procedure.
3. Non-target lesion PCI in the target vessel 24 hours to 30 days.
4. Planned staged procedures.
5. Brachytherapy in conjunction with the index procedure.
6. History of stent thrombosis.
7. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including IABP.
8. Subject is intubated.
9. Known LVEF <30%.
10. Relative or absolute contraindication to DAPT for 6 months in non-ACS patients and 12 months in ACS patients (including planned surgeries that cannot be delayed, or subject is indicated for chronic oral anticoagulant treatment).
11. eGFR <30 mL/min
12. Hemoglobin <10 g/dL.
13. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
14. White blood cell (WBC) count <3,000 cells/mm3.
15. Clinically significant liver disease.
16. Active peptic ulcer or active bleeding from any site.
17. Bleeding from any site within the prior 8 weeks requiring active medical or surgical attention.
18. If femoral access is planned, significant peripheral arterial disease which precludes safe insertion of a 6F sheath.
19. History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
20. Cerebrovascular accident or transient ischemic attack within the past 6 months, or any permanent neurologic defect attributed to CVA.
21. Known allergy to the study stent components cobalt, nickel, chromium, molybdenum, Carbosil®, PBMA, or limus drugs (ridaforolimus, zotarolimus, tacrolimus, sirolimus, everolimus, or similar drugs or any other analogue or derivative or similar compounds).
22. Known allergy to protocol-required concomitant medications such as aspirin, or DAPT (clopidogrel, prasugrel, ticagrelor), or heparin and bivalirudin, or iodinated contrast that cannot be adequately pre-medicated.
23. Any co-morbid condition that may cause non-compliance with the protocol (e.g. dementia, substance abuse, etc.) or reduced life expectancy to <24 months (e.g. cancer, severe heart failure, severe lung disease).
24. Patient is participating in or plans to participate in any other investigational drug or device clinical trial that has not reached its primary endpoint.
25. Women who are pregnant or breastfeeding.
26. Women who intend to become pregnant within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure).
27. Patient has received an organ transplant or is on a waiting list for an organ transplant.
28. Patient is receiving or scheduled to receive chemotherapy within 30 days before or any time after the index procedure.
29. Patient is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease (e.g., HIV). Corticosteroids are allowed.

    Angiographic Exclusion Criteria (visual estimate):
30. Unprotected left main lesions ≥30%, or planned left main intervention.
31. Bifurcation lesions with planned dual stent implantation.
32. Stenting of lesions due to DES restenosis.
33. Occlusive thrombus and/or a thrombus requiring thrombectomy in a target vessel
34. Another lesion in a target or non-target vessel (including all side branches) is present that requires or has a high probability of requiring PCI within 12 months after the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent PCI for angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present), NSTEMI, and recent STEMI (>24 hours from initial presentation and stable) with attempted implantation of a 2.25 mm diameter EluNIR stent.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
MACE | At 30 days
  Combined early efficacy and safety endpoint:
  MACE at 30 days for all patients enrolled. MACE is defined as the composite of cardiac death, any MI, or ischemia-driven TLR.
TLF | At 6 month
  Combined late efficacy and safety endpoint:
  Target Lesion Failure (TLF) at 6 months (evaluated for the first 50% of patients enrolled) Defined as the composite of cardiac death, target vessel-related myocardial infarction, or ischemia-driven target lesion revascularization.

SECONDARY OUTCOMES:
TLF | 6 Months and 1 Year
  Target Lesion Failure at 6 months (for all patients enrolled) and 1 year
Device success | 30 Days, 6 Months & 1 Year
  Device success is defined as achievement of a final in-stent residual diameter stenosis of <30% (by QCA), using the EluNIR 2.25 mm stent only and without a device malfunction.
Lesion success | 30 Days, 6 Months & 1Year
  Lesion success is defined as achievement of a final in-stent residual diameter stenosis of <30% (by QCA) using any percutaneous method.
Procedure success | 30 Days, 6 Months & 1Year
  Procedure success is defined as achievement of a final in-stent diameter stenosis of <30% (by QCA) using the assigned device and/or with any adjunctive devices, without the occurrence of cardiac death, Q wave or non-Q wave MI, or repeat revascularization of the target lesion during the hospital stay.
Target vessel failure | 30 Days, 6 Months & 1 Year
  TVF; the composite rate of death, target vessel related MI or ischemia-driven TVR)
Major adverse cardiac events | 30 Days, 6 Months & 1Year
  MACE; the composite rate of cardiac death, any MI or ischemia-driven TLR
All-cause mortality | 30 Days, 6 Months & 1 Year
  cardiac death, vascular death, non cardiac death
Cardiac death | 30 Days, 6 Months & 1Year
  Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
MI | 30 Days, 6 Months & 1Year
  Post-PCI (Type 4a) and post-CABG (Periprocedural) MIs (Type 5), Periprocedural MIs will be defined based on the SCAI definitions and Spontaneous MI (MI Type I) will be defined based on the Universal Definition of Myocardial Infarction
Target vessel related MI | 30 Days, 6 Months & 1 Year
  Target vessel related MI
Ischemia-driven TLR | 30 Days, 6 Months & 1 Year
  TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion
Ischemia-driven TVR | 30 Days, 6 Months & 1Year
  TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel).
Stent thrombosis | 30 Days, 6Months & 1Year
  ARC definite and probable (Circulation 2007;115:2344-51)

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Richter, PhD, Study Director — Sponsor GmbH
Locations (9):
- Israel (9):
  - Soroka Medical Center, Beersheba
  - Hillel Yafe Medical Center, Hadera
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv